CLINICAL TRIAL: NCT03728114
Title: Effects of Remote Ischemic Conditioning on Cognitive Function and Blood Oxygen Levels in Unacclimatized Adult at High Altitude
Brief Title: Effects of RIC on Cognitive Function and Blood Oxygen Levels in Unacclimatized Adult at High Altitude
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ERIC-HA
Record Dates: First submitted 2018-10-25; First posted 2018-11-01 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Adult
Keywords: adult; remote ischemic conditioning; high altitude condition; cognitive function; blood oxygen levels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High Altitude RIC group (Experimental): Thirty young healthy males from the altitude of 3700 meters will be allocated to the High Altitude RIC group. They will undergo RIC procedure during which bilateral arm cuffs are inflated to a pressure of 200 mmHg for five cycles of 5 min followed by 5 min of relaxation of the cuffs, performed twice a day for a total of 7 days. The treatment was carried out using an electric auto-control device (patent number ZL200820123637.X, China)
  Interventions: Device: RIC
- High Altitude Sham group (Sham Comparator): Thirty young healthy males from the altitude of 3700 meters will be allocated to the High Altitude Sham group. They will undergo a sham RIC procedure during which bilateral arm cuffs are inflated to a pressure of 60 mmHg for five cycles of 5 min, followed by 5 min of relaxation of the cuffs, performed twice a day for a total of 7 days.
  Interventions: Device: sham RIC
- Low Altitude RIC group (Experimental): Thirty young healthy males from the altitude of 42 meters will be allocated to the Low Altitude RIC group. They will undergo RIC procedure during which bilateral arm cuffs are inflated to a pressure of 200 mmHg for five cycles of 5 min followed by 5 min of relaxation of the cuffs, performed twice a day for a total of 7 days. The treatment was carried out using an electric auto-control device.
  Interventions: Device: RIC
- Low Altitude Sham group (Sham Comparator): Thirty young healthy males from the altitude of 42 meters will be allocated to the Low Altitude Sham group. They will undergo a sham RIC procedure during which bilateral arm cuffs are inflated to a pressure of 60 mmHg for five cycles of 5 min, followed by 5 min of relaxation of the cuffs, performed twice a day for a total of 7 days.
  Interventions: Device: sham RIC

INTERVENTIONS:
Device: RIC — Adults allocated to the RIC group will undergo RIC procedure during which bilateral arm cuffs are inflated to a pressure of 200 mmHg over systolic blood pressure for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Arms: High Altitude RIC group; Low Altitude RIC group
Device: sham RIC — Adults allocated to the sham group will undergo a sham RIC procedure during which bilateral arm cuffs are inflated to a pressure of 60 mmHg for five cycles of 5 min, followed by 5 min of relaxation of the cuffs.
  Arms: High Altitude Sham group; Low Altitude Sham group

SUMMARY:
Several studies have shown cognitive impairment such as memory, perception and learning skill during ascent to high altitudes. However, few studies have directly investigated the effect of high altitudes exposure on attention-a high-level cognitive function. Remote ischemic conditioning (RIC) is a noninvasive and easy-to-use neuroprotective strategy, It has been proven to be an effective strategy for neuroprotection in ischemic stroke and chronic cerebral ischemia patients.

DETAILED DESCRIPTION:
This study will provide insights into the preliminary proof of principle, safety, cognitive dysfunction and blood oxygen levels protective effects of RIC in Adults Exposing to High Altitude Conditions, and this data will provide parameters for future larger scale clinical trials if efficacious.

ELIGIBILITY:
Inclusion Criteria:

* The age was between 19 and 30 years.
* All participants should meet the criteria which included right-hand dominance, normal or corrected-to-normal vision.
* the RIC group volunteers have no history of intravascular thrombosis in the bilateral upper limbs;
* The high altitude participants move into the high-altitude environment within one month, and the low altitude volunteers have long-term life in low altitude areas.

Exclusion Criteria:

* Severe hepatic or renal dysfunction
* Severe hemostatic disorder or severe coagulation dysfunction
* Any of the following cardiac disease - rheumatic mitral and or aortic stenosis, prosthetic heart valves, atrial fibrillation, atrial flutter, sick sinus syndrome, left atrial myxoma, patent foramen ovale, left ventricular mural thrombus or valvular vegetation, congestive heart failure, bacterial endocarditis, or any other cardiovascular condition interfering with participation
* Serious, advanced, or terminal illnesses with anticipated life expectancy of less than one year
* Patient participating in a study involving other drug or device trial study 7. Patients with existing neurological or psychiatric disease that would confound the neurological or functional evaluations 8. Unlikely to be available for follow-up for 3 months 9. Contraindication for RIC - severe soft-tissue injury, fracture, or peripheral vascular disease in the upper limbs.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Attentional network test | change from baseline (pre-RIC treatment) at 7days after RIC treatment
  The computer software attentional network test (ANT) as described by Fan et al. in 2002 will be used to measuring the Orienting function, executive function and alerting function.

SECONDARY OUTCOMES:
basic fibroblast growth factor | change from baseline (pre-RIC treatment) at 7 days after RIC treatment
  basic fibroblast growth factor will be detected. Blood samples will be drawn from cubital vein to test these biomarkers.
platelet derived growth factor | change from baseline (pre-RIC treatment) at 7 days after RIC treatment
  platelet derived growth facto will be detected. Blood samples will be drawn from cubital vein to test these biomarkers.
vascular endothelial growth factor | change from baseline (pre-RIC treatment) at 7 days after RIC treatment
  vascular endothelial growth factor will be detected. Blood samples will be drawn from cubital vein to test these biomarkers.
the rate of Adverse event | change from baseline (pre-RIC treatment) at 7 days after RIC treatment
  Any adverse event will be reported and its relationship with the RIC intervention will be evaluated.
distal radial pulses | within 7 days after RIC treatment
  It is an aspect which can reflect the safety of remote ischemic conditioning
the number of erythema in the skin | within 7 days after RIC treatment
  It is an aspect which can reflect the safety of remote ischemic conditioning
the number of patients not tolerating RIC procedure,and refuse to continue the RIC procedure | within 7 days after RIC treatment
  it is an aspect which can reflect the safety of remote ischemic conditioning
the number of patients with any other adverse events related to RIC intervention as determined by the principle investigator. | within 7 days after RIC treatment
  it is an aspect which can reflect the safety of remote ischemic conditioning
heart rate | change from baseline(pre-RIC treatment) at 7days after RIC treatment
  the heart rate will be measured by automatic blood pressure monitor
blood pressure | change from baseline(pre-RIC treatment) at 7days after RIC treatment
  Both systolic, and diastolic pressure will be measured by automatic blood pressure monitor
blood oxygen saturation (SaO2) | change from baseline(pre-RIC treatment) at 7days after RIC treatment
  The portable oxygen saturation ward apparatus (Datex -Ohmeda, USA) will be used to monitor the blood oxygen saturation (SaO2)
cerebral oxygen saturation(TOI) | change from baseline(pre-RIC treatment) at 7days after RIC treatment
  The cerebral oxygen monitor (EGOS-600, Jiangsu China) will be used to monitor the cerebral oxygen saturation (TOI).
The peak systolic blood flow velocity (PSV) of bilateral middle cerebral artery (MCA) | change from baseline(pre-RIC treatment) at 7days after RIC treatment
  This is a indicator of hemodynamic data ,it is measured by Transcranial Doppler ((DWL Doppler-Box, German) according to applicational specifications and technical standards
end-diastolic blood flow velocity (EDV) of bilateral middle cerebral artery (MCA) | change from baseline(pre-RIC treatment) at 7days after RIC treatment
  This is a indicator of hemodynamic data ,it is measured by Transcranial Doppler ((DWL Doppler-Box, German) according to applicational specifications and technical standards
the mean flow velocity (MFV) of the subjects' bilateral middle cerebral artery (MCA) | change from baseline (pre-RIC treatment) at 7 days after RIC treatment
  This is a indicator of hemodynamic data ,it is measured by Transcranial Doppler ((DWL Doppler-Box, German) according to applicational specifications and technical standards
pulse index (PI) of the subjects' bilateral middle cerebral artery (MCA) | change from baseline (pre-RIC treatment) at 7 days after RIC treatment
  This is a indicator of hemodynamic data ,it is measured by Transcranial Doppler ((DWL Doppler-Box, German) according to applicational specifications and technical standards
The degree of palpation of tenderness--visual analogue scale | within 7 days after RIC treatment
  The degree of palpation of tenderness is an aspect which can reflect the safety of remote ischemic conditioning. The pain was assessed with visual analogue scale ( VAS)
the number of patients with any other adverse events related to RIC intervention as determined by the principle investigator | within 7 days after RIC treatment
  it is an aspect which can reflect the safety of remote ischemic conditioning

CONTACTS AND LOCATIONS:
Overall Officials: Lian Duan, MD PHD, Study Chair — The 307th Hospital of Military Chinese People's Liberation Army

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wilson MH, Newman S, Imray CH. The cerebral effects of ascent to high altitudes. Lancet Neurol. 2009 Feb;8(2):175-91. doi: 10.1016/S1474-4422(09)70014-6. PMID 19161909
- [Background] Meng R, Asmaro K, Meng L, Liu Y, Ma C, Xi C, Li G, Ren C, Luo Y, Ling F, Jia J, Hua Y, Wang X, Ding Y, Lo EH, Ji X. Upper limb ischemic preconditioning prevents recurrent stroke in intracranial arterial stenosis. Neurology. 2012 Oct 30;79(18):1853-61. doi: 10.1212/WNL.0b013e318271f76a. Epub 2012 Oct 3. PMID 23035060
- [Background] Meng R, Ding Y, Asmaro K, Brogan D, Meng L, Sui M, Shi J, Duan Y, Sun Z, Yu Y, Jia J, Ji X. Ischemic Conditioning Is Safe and Effective for Octo- and Nonagenarians in Stroke Prevention and Treatment. Neurotherapeutics. 2015 Jul;12(3):667-77. doi: 10.1007/s13311-015-0358-6. PMID 25956401
- [Background] Fan J, McCandliss BD, Sommer T, Raz A, Posner MI. Testing the efficiency and independence of attentional networks. J Cogn Neurosci. 2002 Apr 1;14(3):340-7. doi: 10.1162/089892902317361886. PMID 11970796
- [Background] Posner MI, Petersen SE. The attention system of the human brain. Annu Rev Neurosci. 1990;13:25-42. doi: 10.1146/annurev.ne.13.030190.000325. No abstract available. PMID 2183676
- [Background] Godfrey E, Chalder T, Ridsdale L, Seed P, Ogden J. Investigating the active ingredients of cognitive behaviour therapy and counselling for patients with chronic fatigue in primary care: developing a new process measure to assess treatment fidelity and predict outcome. Br J Clin Psychol. 2007 Sep;46(Pt 3):253-72. doi: 10.1348/014466506X147420. PMID 17697477
- [Background] Wang Y, Meng R, Song H, Liu G, Hua Y, Cui D, Zheng L, Feng W, Liebeskind DS, Fisher M, Ji X. Remote Ischemic Conditioning May Improve Outcomes of Patients With Cerebral Small-Vessel Disease. Stroke. 2017 Nov;48(11):3064-3072. doi: 10.1161/STROKEAHA.117.017691. Epub 2017 Oct 17. PMID 29042490
- [Background] Twomey R, Wrightson J, Fletcher H, Avraam S, Ross E, Dekerle J. Exercise-induced Fatigue in Severe Hypoxia after an Intermittent Hypoxic Protocol. Med Sci Sports Exerc. 2017 Dec;49(12):2422-2432. doi: 10.1249/MSS.0000000000001371. PMID 28708702